# Acne Research Studies – Assessing Eligibility for Clinical Trial Participation

The Informed Consent Process in <a href="Power Clinical Trial's">Power Clinical Trial's</a>
Observational Study: A Guide for Participants

Date: May 30, 2025

The Informed Consent Document Explained

If you are asked to fill out this form, this means you are being considered for participation in an observational clinical trial focused on patients with acne.

It outlines the study in detail, including its goals, implementation, and both the positive and negative aspects. It is important to weigh your options before deciding to participate and to reach out to someone you trust for their input.

If there are any misunderstandings or questions about the information contained in this document, feel free to approach the researcher for clarification.

The Aim of the Clinical Trial for Acne

Acne is a common skin condition characterized by the appearance of pimples, blackheads, and whiteheads. It occurs when hair follicles become clogged with oil and dead skin cells, leading to the growth of bacteria in the area and causing inflammation.

Acne clinical trials are conducted to test the safety and efficacy of new treatments for acne. These trials are necessary to determine whether new treatments are better than existing ones and to provide evidence that supports the use of these treatments in the general population.

The purpose of this study is to scrutinize the experiences of patients diagnosed with acne as they take part in a separate medical intervention clinical trial. The focus will be on tracking the rates of completion and withdrawal among these individuals.

## Understanding the Nature of an Observational Clinical Trial

As a participant in this medical trial, you will be a part of an observational study, which is a type of clinical trial that aims to gather information by observing individuals without making any changes to their care plans.

Researchers will simply observe you and measure the outcomes of the condition without intervening in any way. This type of trial is an important tool for gaining a deeper understanding of the natural progression of a particular condition, and the effects it has on individuals who are diagnosed with it.

By participating in this observational study, you will be contributing to the advancement of medical knowledge and helping to improve the care of individuals who have the same condition.

## More Acne Clinical Trials Comparison

This clinical trial is observational, meaning that you will not be receiving any specific treatments or interventions as a part of the study. However, there are many other types of clinical trials for acne that are interventional in nature and require participants to undergo a specific treatment.

To make an informed decision about whether you would like to participate in a clinical trial, it's important to research and compare different studies. You can access information about <u>acne studies</u> by visiting clinicaltrials.gov or checking out Power's website, which offers <u>acne clinical trials</u> that are open for recruitment.

By taking the time to research and understand the different types of clinical trials available, you can make a well-informed decision about whether participation in a trial is right for you.

## Voluntary Participation in Clinical Trial Surveys

As a participant in this observational clinical trial, we would like to gather information about your experiences. This will be done through the completion of questionnaires every two weeks, which should take approximately 20-30 minutes. In addition, we will conduct check-in calls on a quarterly basis for as long as you continue to participate in the trial.

It's important to emphasize that your participation in the survey aspect of the trial is completely optional. You are not required to answer any or all questions, and you have the right to terminate your involvement in the trial at any time if you so choose. We understand that participating in a clinical trial can be a personal decision, and we are committed to supporting you in any way we can. Your privacy and comfort are of the utmost importance to us, and we will respect your decision-making process throughout the trial.

## Anonymity of Responses

The confidentiality of your information is a top priority during this clinical trial. To ensure your anonymity, kindly refrain from providing any personal or identifying details in your answers to the questionnaires.

The research team will take every step to safeguard your confidentiality. Nonetheless, there may be specific legal situations in which the researcher is required to share your data.

#### **Benefits**

Participating in this observational clinical trial will not provide immediate benefits for individuals, but their contribution can make a lasting impact on the lives of others.

The data gathered from the participants will be used to improve the enrolment process for future acne patients, making it easier for them to access medical research opportunities. By joining this clinical trial, individuals will have the opportunity to make a difference for future acne patients and contribute to the advancement of medical research.

#### Risks

Clinical trials have been instrumental in advancing the medical field, but they can also pose health risks to participants, especially when receiving novel treatments.

However, our observational clinical trial eliminates this risk by not requiring participants to receive any new interventions. Instead, participants are observed, and outcomes are measured, without exposing them to any unnecessary health risks.

The confidentiality of participant information is a significant concern in clinical trials. Our medical study has taken several steps to ensure the privacy of participant data. All data collected from participants are anonymous, and access to this information is restricted to the research team only.

Furthermore, all records, including call logs, online transactions, forms, and surveys, are stored securely with encryption and password protection. This ensures that participant information remains confidential and protected from unauthorized access.

# Voluntary Participation in the Acne Clinical Trial

Your participation in the acne clinical trial is voluntary. It is entirely up to you to decide whether or not you will join this study. If you join, you will need to sign this informed consent form. After you sign this document, you are still free to stop your participation at any time and even without giving any reason.

# Additional Research on Clinical Trial Diversity

For those who want to dive deeper into the topic of representation in clinical trials, there are a wealth of online resources available.

Whether you're looking to gain a better understanding of the challenges and opportunities, or simply seeking information to inform your involvement in clinical trials, these resources can be an invaluable resource:

Polo, Antonio J., Bridget A. Makol, Ashley S. Castro, Nicole Colón-Quintana, Amanda E. Wagstaff, and Sisi Guo. "Diversity in randomized clinical trials of depression: A 36-year review." *Clinical Psychology Review* 67 (2019): 22-35.

Lindenfeld, JoAnn, Mona Fiuzat, and Christopher O'Connor. "Promoting diversity in clinical trial leadership: a call to action." *Heart Failure* 9, no. 5 (2021): 401-402.

## **Statement Providing Consent**

I affirm that I have taken the time to thoroughly read and comprehend the informed consent form, either independently or with the aid of a trusted individual who has read it to me. All my questions and concerns have been addressed to my satisfaction.

I fully understand that my participation in this study is entirely voluntary and that I have the right to withdraw my consent at any moment, without having to provide a reason or incur any fees. I have been informed that a copy of this informed consent form will be provided to me for my records.

After careful consideration and weighing of all the information presented to me, I agree to participate in this study of my own free will.

| Printed Name of Participant |
|-----------------------------|
| Participant Signature |
| <br>Date |

## **Declaration of Person Taking Consent**

I have thoroughly reviewed the information contained in this document with the participant, ensuring that they have a clear understanding of the purpose, methods, potential risks and benefits, and other crucial aspects of the acne clinical trial.

The participant was provided ample opportunity to ask questions and have any confusion or misunderstandings addressed. It is important to note that their participation in this trial is completely voluntary and they are free to withdraw at any time, for any reason, without incurring any costs.

Upon providing their consent, a copy of this document was provided to the participant for their records.

| Printed Name of Person Taking Consent |
|---------------------------------------|
| Signature of Person Taking Consent |
| <br>Date |